CLINICAL TRIAL: NCT00629993
Title: Dissemination of Cervical Cancer Screening to Primary Care Physicians in Underserved Communities
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal Investigator left the institution
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Vicki Benard, Ph.D., Project Officer, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: AAAA9722; U57/CCU224079
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer screening; medically underserved women; HPV vaccine
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multi-component Academic Detailing (Experimental): Multi-component, academic detailing regarding ACS guidelines on cervical cancer screening approaches.
  Includes an interactive, digitized CD-ROM, focused on the discussion of risks and benefits, screening options or alternatives, values clarification, and mutual decision-making, alongside patient education materials designed for low literacy patients.
  Interventions: Behavioral: Academic Detailing

INTERVENTIONS:
Behavioral: Academic Detailing — It will involve multiple intervention components, some of which are standardized across physicians (i.e., self learning packets, post-tests for CME credit, CD-ROMS, videos, newsletters, culturally sensitive patient education materials, office staff informational sessions, chart and patient reminders, and a general office routine for cervical cancer counseling, including performance feedback, as well as media-ready materials). Academic detailing and the specific office routines will be customized to each physician, although the frequency of the detailing visits will be routinized across all participants, to reduce cost and to maximize its potential for dissemination.
  Other Names: Multi-component Academic Detailing

SUMMARY:
Primary care physicians have an important role to play in the delivery of cancer prevention and detection services to patients. Face-to-face counseling of physicians, called academic detailing, involves a brief and focused intervention, modeled on the practices of pharmaceutical companies. This type of intervention may increase physicians' attention to preventive opportunities and increase their screening behaviors.

DETAILED DESCRIPTION:
The specific aims of this proposal are:

1. To test the hypothesis that an intervention, multi-component academic detailing, will increase the rate of physician cervical cancer screening at 3- and 6-months post-randomization, compared to the rate observed in a service-as-usual control.
2. To develop models predicting which physician offices are most and least likely to adopt the intervention, and to generate hypotheses about tailoring the dissemination of cervical cancer screening guidelines to different physician subgroups.
3. To conduct a cost-effectiveness analysis comparing the incremental societal costs and effects (in lives saved, life-years saved, and quality-of-life-years saved) of the cervical cancer intervention implemented in physicians' offices.

The long-term goal of this project therefore is to reduce cervical cancer risks among ethnic and racial minorities, by influencing the screening behaviors of their primary care physicians.

ELIGIBILITY:
Inclusion Criteria:

* Charts of female patients age 18-85 with at least one visit to the primary care provider over the last two years will be reviewed

Exclusion Criteria:

* Exclusion criteria will include: diagnosis of cancer other than non-melanotic skin cancer and removal of the uterus.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2004-01; Primary Completion 2006-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Number of asymptomatic female patients age 18-85 who receive or are referred for a recto-pelvic bimanual examination with the collection of the Pap smear (per ACS guidelines); collected via medical chart review | 12-month followup

SECONDARY OUTCOMES:
Physician knowledge, attitudes and beliefs toward cervical cancer prevention, screening, and treatment | 12-month followup

CONTACTS AND LOCATIONS:
Overall Officials: Sherri Sheinfeld Gorin, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States